CLINICAL TRIAL: NCT03471728
Title: [PMS] LINZESS® Tablet 0.25mg Long-term Specified Drug Use-results Survey in Patients With Irritable Bowel Syndrome With Constipation or Chronic Constipation (Excluding Constipation Due to Organic Diseases)
Brief Title: Post-marketing Surveillance of Linaclotide Tablet in Patients With Irritable Bowel Syndrome With Constipation or Chronic Constipation (Excluding Constipation Due to Organic Diseases)
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: 0456-MA-3141
Record Dates: First submitted 2018-03-14; First posted 2018-03-21 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Chronic Constipation (CC) (Excluding Constipation Due to Organic Diseases); Irritable Bowel Syndrome With Constipation (IBS-C)
Keywords: Linaclotide; Linzess; Irritable Bowel Syndrome; Chronic Constipation
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — linaclotide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Irritable Bowel Syndrome: Patients with Irritable Bowel Syndrome with Constipation (IBS-C) who have used linaclotide for the first time
  Interventions: Drug: linaclotide
- Chronic Constipation: Patients with Chronic Constipation (CC) (excluding constipation due to organic diseases) who have used linaclotide for the first time
  Interventions: Drug: linaclotide

INTERVENTIONS:
Drug: linaclotide — Oral
  Other Names: Linzess; ASP0456

SUMMARY:
The objective of this study is to evaluate the long-term safety and efficacy of linaclotide in post-marketing use.

DETAILED DESCRIPTION:
This is a post-marketing long-term specified drug use-result survey study required for products in Japan. The investigator will register the patient who have been taking this product for the first time within 14 days after the start of treatment (inclusive of the start day). For each of the registered patients (including withdrawals and dropouts), the investigator will enter the survey data on the case report form.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Irritable Bowel Syndrome with Constipation (IBS-C) or Chronic Constipation (CC) (excluding constipation due to organic diseases) who have used linaclotide for the first time

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Irritable Bowel Syndrome with Constipation (IBS-C) or Chronic Constipation (CC) (excluding constipation due to organic diseases) who have used linaclotide for the first time
Sampling Method: Non-Probability Sample
Enrollment: 2475 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of diarrhea | Up to Week 36
  To assess the incidence of diarrhea as a criteria of safety variables.

SECONDARY OUTCOMES:
Safety assessed by incidence of adverse drug reactions | Up to Week 36
  Adverse drug reactions will be coded using Medical Dictionary for Regulatory Activities (MedDRA).
Efficacy assessed by Global assessment of relief of IBS and constipation symptoms | Up to Week 36
  Global assessment of relief of IBS and constipation symptoms will be evaluated based on the clinical course in a medical interview with the patient and evaluate efficacy using a 7-point scale: 1: much better; 2: better; 3: a little better; 4: no change; 5: a little worse; 6: worse; 7: much worse. If the evaluation is impossible, a reason will be provided.

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Director — Astellas Pharma Inc
Locations (47):
- Japan (47):
  - Site JP00023, Aichi
  - Site JP00005, Akita
  - Site JP00002, Aomori
  - Site JP00012, Chiba
  - Site JP00038, Ehime
  - Site JP00018, Fukui
  - Site JP00040, Fukuoka
  - Site JP00007, Fukushima
  - Site JP00021, Gifu
  - Site JP00010, Gunma
  - Site JP00034, Hiroshima
  - Site JP00001, Hokkaido
  - Site JP00028, Hyōgo
  - Site JP00008, Ibaraki
  - Site JP00017, Ishikawa
  - Site JP00037, Kagawa
  - Site JP00046, Kagoshima
  - Site JP00014, Kanagawa
  - Site JP00039, Kochi
  - Site JP00043, Kumamoto
  - Site JP00026, Kyoto
  - Site JP00024, Mie
  - Site JP00004, Miyagi
  - Site JP00045, Miyazaki
  - Site JP00020, Nagano
  - Site JP00042, Nagasaki
  - Site JP00029, Nara
  - Site JP00015, Niigata
  - Site JP00003, Numakunai
  - Site JP00033, Okayama
  - Site JP00047, Okinawa
  - Site JP00027, Osaka
  - Site JP00044, Ōita
  - Site JP00041, Saga
  - Site JP00011, Saitama
  - Site JP00025, Shiga
  - Site JP00032, Shimane
  - Site JP00022, Shizuoka
  - Site JP00009, Tochigi
  - Site JP00036, Tokushima
  - Site JP00013, Tokyo
  - Site JP00031, Tottori
  - Site JP00016, Toyama
  - Site JP00030, Wakayama
  - Site JP00006, Yamagata
  - Site JP00035, Yamaguchi
  - Site JP00019, Yamanashi

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.